CLINICAL TRIAL: NCT05017129
Title: E-training of Inmate Peer Caregivers for Enhancing Geriatric and End-of-life Care in Prisons - Phase II
Brief Title: E-training of Inmate Peer Caregivers for Enhancing Geriatric and End-of-life Care in Prisons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Penn State University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0327; 5R44AG057239-03 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2021-08-23 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: Cognitive interviews and small-scale usability will be conducted prior to conducting the full-scale testing. The full-scale learning system (6 learning modules for inmates; 1 learning module for staff) will be tested in 12 state prison settings. We plan to use a pragmatic approach. Targeted participants to test the inmate-focused modules will include both current Inmate Peer Caregivers and inmates who are naïve to the caregiving role in prison. Staff participants to test the staff-focused module include, but are not limited to security, chaplaincy, medical services, psychology/counseling, and administrative leaders. The number of user-participants is dependent on the institution's size, but our target is to recruit 12 sites (three of which will be women's prisons) and an average of 20 inmates per site (n=240 inmates) to test the six modules that are developed for inmates and an average of four prison staff per site (n=48) to test the one module for staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inmates Care modules (Experimental): This is a within-subjects, pre-post design with a single intervention. The intervention is a 6 module computer-based learning program for training peer caregivers in end-of-life care.
  Interventions: Behavioral: Inmates Care

INTERVENTIONS:
Behavioral: Inmates Care — The single intervention is a computer-based learning program.

SUMMARY:
The demographics of the U.S. prison population are shifting at a dramatic rate requiring new approaches to prison healthcare. Current estimates suggest that there are 2.3 million incarcerated persons in the U.S. Similar to the free world, the aging of the Baby Boom generation is occurring in prisons. Notably, inmates 50 and older constitute over 20% of prisoners in state or federal facilities. From 1996-2016, there was an 280% growth in the number of state and federal prisoners age 55 or older, which is in sharp contrast to younger inmates that grew by only 3% during this time period. A surge in older adult offenders in the U.S. has not occurred but rather statutes now impose stiffer sentences, resulting in longer periods of incarceration, such as life without parole or 20+ years. At the same time, early release policies remain restrictive. As a result, sentenced offenders are living through middle and older adulthood within the confines of prisons.

DETAILED DESCRIPTION:
There are over 1,719 United States (US) state and federal prisons with over 2.3 million prisoners. In 2017, more than 20% of sentenced prisoners were age 50 or older. The health status of older inmates is often parallel with free-living people who are far older (e.g., 10-15 years). Older prisoners disproportionately contribute to the steeply rising correctional healthcare costs and their death rate is 10 times that of younger prisoners. Corrections budgets are stretched as they strive to meet the care needs of aged and dying prisoners. Carefully selected and vetted inmates offer an abundant human resource that is poised to contribute in important ways to augment prison staff in meeting growing care needs of older and dying inmates. However, the lack of standardized, evidence-based, training that is geared toward this target audience is a current barrier to ensuring high quality inmate caregiving. In response to this need, our Phase I project E-training of Inmate Peer Caregivers for Enhancing Geriatric and End-of-Life Care in Prisons demonstrated that inmate access to technology is growing and inmates can be successful e-learners. Specifically, we learned: (1) there is a need and interest for products such as our Inmates Care computer-based learning (CBL); (2) trainings should be engaging, interactive, and contextually sensitive to the specific environment, target user, and security constraints, while at the same time being mindful of emerging trends in regard to technology use by inmates (e.g., availability of tablets for purchase and use in many states); and finally, (3) that interactive, media-rich prototype modules with high acceptability and usability could be developed. The specifications document and commercialization plan indicated it is possible to develop a full-scale Inmates Care learning system in Phase II and a Technology Niche Analyses® revealed market potential exists. The purpose of this Phase II application is to continue research and development of the Inmates Care learning system with an emphasis on developing a scalable unit for commercialization and testing scale-up in a larger number of more diverse state prisons. More specifically, the aims of this Phase II study are to: 1) Develop a full scale media-rich interactive computer-based learning system Inmates Care, that consists of six modules aimed at augmenting the highly variable face-to-face inmate caregiving programs in state prisons with standardized, evidence-based training to prepare inmates in assisting with end-of-life (EOL) and geriatric care; and one Training Overview and Rollout module that prepares staff to use Inmates Care as a tool for inmate peer caregiver training; 2) Conduct in-person usability testing of the full-scale Inmates Care program in two rounds in state prisons to evaluate logistics, inmate and staff impressions, user interface, ease of use, and perceived barriers in order to optimize the scalable unit for broader dissemination (n=30); and 3) Test scale-up of the full-scale Inmates Care program in state prisons across the nation to evaluate knowledge acquisition outcomes, usage patterns, and commercialization opportunities (n=288).

ELIGIBILITY:
Inclusion Criteria:

Inmate Peer Caregivers:

1. providing geriatric and/or EOL care at participating state prison (Aims 1 and 2 only);
2. age >18;
3. able to speak and understand English; and
4. able to consent.

Exclusion Criteria:

1. Under the age of 18
2. Unable to speak and understand English

Prison Staff:

Inclusion Criteria:

1. age >18;
2. able to speak and understand English;
3. able to consent; and
4. have been exposed to inmate peer caregiving (e.g., through training them, oversight of a peer caregiving program, or working with inmate peer caregivers in the infirmary, personal care, or hospice area of prisons)

Exclusion Criteria:

1. Under the age of 18
2. Unable to speak and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge Acquisition | Pre-test (prior to online training- Total Score)
  There are no existing measures to evaluate improvements in knowledge among inmates and staff for geriatric and EOL care of inmates. Therefore, the primary outcome measure will be developed for this project. Scale development and psychometric properties will be evaluated (e.g., content-validity, criterion-related validity, construct validity, and internal consistency) using: (1) domain identification and item generation; (2) content expert validation, and (3) pilot test.
Inmates Program Findings | Post-test (immediately following online training) approximately one hour
  Evaluate improvements in knowledge among inmates

SECONDARY OUTCOMES:
System Usability Scale (SUS) | After small-scale usability testing and at post-test for the large-scale testing. Approximately two hours
  The SUS is a validated tool for assessing the usability and acceptability of technological products.
Qualitative questions | After small-scale usability testing and at post-test for the large-scale testing. Approximately two hours
  Six brief open-end questions that ask how helpful the program was, how the liked program was, and whether the user has any suggested changes to the program.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Walkosz, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Klein Buendel, Inc., Golden, Colorado
  - Pennsylvania State University, University Park, Pennsylvania

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT05017129/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT05017129/ICF_001.pdf